CLINICAL TRIAL: NCT05243914
Title: Heart Transplantation Using Normothermic Regional Perfusion (NRP) Donation After Circulatory Death (DCD): A Pilot Study
Brief Title: Heart Transplantation Utilizing NRP DCD
Status: Terminated | Type: Observational
Why Stopped: Slow study enrollment
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Radha Gopalan, Clinical Assistant Professor, Internal Medicine, University of Arizona
Other Study IDs: STUDY00000230
Record Dates: First submitted 2022-01-21; First posted 2022-02-17 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Heart Transplantation; Perfusion; Transplant Recipients
Keywords: Normothermic Regional Perfusion (NRP); Donation After Circulatory Death (DCD); Heart Transplantation; Observational Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, observational, pilot trial to evaluate the feasibility of heart transplantation using normothermic regional perfusion (NRP) donation after donor circulatory death (DCD). Adults who meet standard criteria for heart transplantation listing and study-specific eligibility criteria will enroll in the study.

the investigators anticipate evaluating an initial cohort of approximately 100 DCD donors for a final yield of 40 hearts. The investigators will accept donors between the ages of 18 and 65 who are determined to have heart function/quality appropriate for donation for transplantation based on available donor data and testing.

If feasible, donors might be relocated to BUMCP to maintain uniformity of process, minimize cold ischemic time, and allow for more rapid and improved communication during the initial pilot phase.

Recipients will be selected based on blood group, crossmatch, size match, and clinical stability per standard allocation practices. Recipients will be followed post-transplantation per BUMCP Heart Transplant standard protocol.

DETAILED DESCRIPTION:
The surgical management of end-stage heart failure generally falls into two categories: mechanical circulatory support and heart transplantation. The availability of suitable organs intrinsically limits the rate of heart transplantation. The vast majority of cadaveric donor hearts are obtained from patients who have had irreversible cessation of neurological function (DBD - Donation after Brain Death). Recently, there has been renewed interest in the possibility of obtaining cadaveric hearts from DCD (Donation after Circulatory Death) donors who have had irreversible cessation of cardiopulmonary function. In contrast to DBD, DCD involves the intentional withdrawal of life support measures to allow controlled circulatory death to occur. If the patient fails to progress to circulatory death within the allotted time, DCD donation is terminated, and the patient is placed on comfort measures until they expire.

The concept of DCD heart transplantation is not new. Barnard used DCD hearts in his early series of heart transplants because the idea of brain death had not yet been well established. Clinical DCD heart transplant programs have been established in the UK, Belgium, and Australia. However, DCD heart transplantation currently remains virtually nonexistent in the US. DCD can increase the available US heart donor pool by as much as 20%. Of the more than 41,000 adult heart transplants performed in the US over the past 20 years, only 4 have been from DCD donors. Perhaps understandably, there is some hesitance in using a donor heart that has just undergone circulatory death.

Potential DCD donors are stratified according to the Maastricht classification system: 1) dead on arrival at the hospital, 2) out-of-hospital arrest with unsuccessful resuscitation, 3) circulatory arrest as a result of a planned withdrawal of life support, 4) circulatory arrest in a patient who is already brain-dead, and 5) circulatory arrest while in the hospital with unsuccessful resuscitation. Categories 1, 2, and 5 would be considered "uncontrolled" DCD. Categories 3 and 4 are considered "controlled" DCD, where the duration and conditions of warm ischemia are known, and the precise course of circulatory arrest can be followed.

The current procedure of DCD organ donation and procurement follows a well-established course for lung, liver, kidney, and pancreas transplantation in the United States. After consent has been obtained, the organs are allocated through the United Network of Organ Sharing (UNOS). When all parties are present and ready, the donor is withdrawn from life support (i.e., discontinuation of mechanical ventilation and any vasoactive medications). The surgical teams are generally present on the premises but not at the donor's bedside. After circulatory arrest occurs, which is determined by the absence of pulse and organized rhythmic cardiac activity, death is declared by a physician not associated with the transplant teams. Subsequently, a standoff period is observed (5 minutes) to ensure a complete cessation of the circulation before organ procurement is commenced. If after withdrawal of life support, the patient does not progress to circulatory death within the allotted time (variable among hospitals, but 60 minutes in this study), the procurement is abandoned, and the patient is transferred out of the operating room and placed on palliative measures.

Given that DCD organ donation is already currently practiced in the US, the same standard approach defined by each state and locality can also be applied to DCD heart donation. However, this protocol will utilize a normothermic regional perfusion (NRP) strategy that involves the re-establishment of circulatory blood flow after the period of circulatory arrest has been established and the 5 minutes of standoff time has passed. The local Organ Procurement Organization (Donor Network of Arizona-DNAZ) and BUMCP Leadership have reviewed and approved this approach to DCD heart donation. Specifically, normothermic regional perfusion involves the following steps:

1. Opening the chest through a standard sternotomy used for heart and lung procurement.
2. Ligation of all the blood vessels that supply blood to the brain to ensure that blood flow to the brain is not re-established once circulation is restarted, as described below.
3. Standard cannulation of the aorta and the right atrium as is done for cardiac surgical procedures.
4. Initiation of cardiopulmonary bypass, which will re-establish blood flow to all organs of the body, including the heart under normothermia. The initial step for ligation of the blood vessels to the head is necessary to ensure that blood flow to the brain does not occur.

Once blood flow to the heart is established, the heart will start beating. At 30 to 60-minute intervals, the donor will be separated from cardiopulmonary bypass, and the heart will be assessed for functionality. If accepted, standard DBD procurement will commence. The heart transplantation surgery on the potential recipient will only begin once the heart has been accepted as suitable.

If, after assessment, the heart is not suitable, cardiopulmonary bypass will be restarted. The donor heart will be reassessed at 30-minute intervals up to 180 minutes. If no significant acceptable recovery occurs and the heart is not deemed suitable for transplantation, then the study will be terminated, but the remaining organs can be recovered as standard practice.

Although there has been limited experience with DCD heart donation in the US up to this point, they are being performed with increasing frequency in Europe and Australia. Although protocols already exist for DCD donation for other organs, there is currently no established US consensus for DCD hearts.

To date researchers have found comparable short-term and midterm results between the standard and DCD heart transplantation techniques, however the longer-term results are unknown at this time. This study will help us learn more about the long-term outcomes and see how well the DCD technique works for heart transplant.

Although the investigators report comparable short-term and midterm results between DBD and DCD heart transplantation, the longer-term results are unknown Regardless of the retrieval protocol utilized, there is now sufficient accumulated clinical experience to indicate that heart transplants from selected DCD donors are associated with outcomes comparable to those observed with DBD donors.

ELIGIBILITY:
Inclusion Criteria:

* Recipient Inclusion Criteria
* Recipient is ≥ 18 years old
* Recipient, or their designated healthcare proxy, is able and willing to sign an informed consent
* The recipient meets standard listing criteria for heart transplantation.

Exclusion Criteria:

* Recipient is < 18 years old
* Recipient, or their designated healthcare proxy, is unable to sign an informed consent
* The recipient is participating in another interventional trial
* The recipient has a known history of HIV infection
* The recipient has any condition that, in the opinion of the Investigator, would make study participation unsafe or would interfere with the objectives of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We anticipate evaluating an initial cohort of approximately 100 DCD donors for a final yield of 40 hearts suitable for transplantation. Donors will be between the ages of 18 and 65 who are determined to have heart function/quality that is appropriate for donation for transplantation based on available donor data and testing. Donors might be transported to BUMCP with the intent of implanting the recipients at BUMCP. It is preferable to relocate the donor and recipient to maintain uniformity of process, minimize cold ischemic time and allow for rapid and improved communication during the initial pilot phase.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of feasibility | through study completion, an average of 1 year
  To evaluate the survival of heart transplantation recipients using normothermic regional perfusion (NRP) donation after circulatory death (DCD).

SECONDARY OUTCOMES:
Evaluation of Incidence of Rejection | through study completion, an average of 1 year
  To evaluate incidence of rejection over an extended period of pump-assisted reperfusion for DCD heart donation.

CONTACTS AND LOCATIONS:
Locations (1):
- Banner University Medical Center Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Data collected for this study will be analyzed and stored in a HIPAA compliant REDCap database hosted by UA. After the study is complete, the de-identified, archived data will be retained in REDCap per the UA IRB guidelines.
  When the study is complete, access to study data will be provided through REDCap. This study will adhere to the UA policy for data sharing.